CLINICAL TRIAL: NCT03213912
Title: Determination of EC50 of Anesthetics During Microelectric Recording in Patients Receiving Deep Brain Stimulation Under Anesthesia
Brief Title: EC50 of Anesthetics During Microelectric Recording
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator, Associate Professor, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2015-12-004B
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Deep Brain Stimulation
Keywords: effective concentration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators determine the half maximum effective concentration (EC50) of the Cet value of propofol in target-controlled infusion (TCI) when co-administered with dexmedetomidine for the maintenance of general anesthesia during microelectrode recording in the deep brain surgery in patients with Parkinson's disease.

DETAILED DESCRIPTION:
General anesthesia is sometimes required for DBS (deep brain stimulation) surgery in those with excessive fear, anxiety, reduced cooperation, or severe movements due to ' off drug' state. Dexmedetomidine and propofol are both used individually in the sedation for DBS surgery, and were reported to affect the MER (microelectrode recording) to some extent, especially in the higher zone of the dose range. In this study, the investigators plan to use the combination of dexmedetomidine and propofol for the maintenance of general anesthesia in patients with Parkinson's disease. In this study, dexmedetomidine is given with a loading dose of 0.5 mcg/Kg, and continuous infusion with the dose of 0.4 mcg/Kg/hr. Propofol is given within 0.8~1.8 mcg/Kg during the MER recording (based on institutional guideline). MER recording will be observed and correlated wtih the dose of propofol. The Dixon "up-and-down" sequential allocation method was used to determine the EC50 of the value of Cet of propofol. The study aims to determine the dose that is adequate for maintaining general anesthesia with endotracheal intubation and least interference with the MER recording.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-85
2. Clinical diagnosis of Parkinson's disease
3. Scheduled for deep brain stimulation surgery under general anesthesia

Exclusion Criteria:

1. Allergic history to dexmedetomidine and propofol
2. Clinical diagnosis of congestive heart failure
3. Clinical diagnosis of liver cirrhosis
4. Clinical diagnosis of third degree A-V block

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, aged 20-85, with clinical diagnosis of Parkinson's disease, who are undergoing deep brain stimulation for which gnenral anesthesia with endotracheal intubation is required.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Cet of propofol | Intraoperative
  concentration of propofol used during microelectrode recording

CONTACTS AND LOCATIONS:
Overall Officials: WT Change, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided